CLINICAL TRIAL: NCT01187199
Title: Phase I Trial of Bevacizumab and Temsirolimus in Combination With 1) Carboplatin, 2) Paclitaxel, 3) Sorafenib for the Treatment of Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0486; NCI-2012-01788 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer
Keywords: Metastatic cancer; Chemotherapy; Avastin; Carboplatin; Paclitaxel; Sorafenib; Temsirolimus
MeSH Terms: conditions — Neoplasm Metastasis | interventions — temsirolimus; Bevacizumab; Paclitaxel; Sorafenib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Carboplatin Group (Experimental): Carboplatin: Starting dose AUC 2 by vein on day 1 of a 21 day cycle. Temsirolimus: Starting dose 12.5 mg by vein given on day 1, 8, and 15 of a 21 day cycle. Bevacizumab: Starting dose 5 mg/kg given by vein on day 1 of a 21 day cycle.
  Interventions: Drug: Temsirolimus; Drug: Bevacizumab; Drug: Carboplatin
- Paclitaxel Group (Experimental): Paclitaxel: Starting dose 30 mg/m2 given by vein on day 1 of a 21 day cycle. Temsirolimus: Starting dose 12.5 mg by vein given on day 1, 8, and 15 of a 21 day cycle. Bevacizumab: Starting dose 5 mg/kg given by vein on day 1 of a 21 day cycle.
  Interventions: Drug: Temsirolimus; Drug: Bevacizumab; Drug: Paclitaxel
- Sorafenib Group (Experimental): Sorafenib: Starting dose 200 mg by mouth daily for a 21 day cycle. Temsirolimus: Starting dose 12.5 mg by vein given on day 1, 8, and 15 of a 21 day cycle. Bevacizumab: Starting dose 5 mg/kg given by vein on day 1 of a 21 day cycle.
  Interventions: Drug: Temsirolimus; Drug: Bevacizumab; Drug: Sorafenib

INTERVENTIONS:
Drug: Temsirolimus — Starting dose 12.5 mg by vein given on day 1, 8, and 15 of a 21 day cycle.
  Other Names: CCI-779; Torisel
Drug: Bevacizumab — Starting dose 5 mg/kg given by vein on day 1 of a 21 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Paclitaxel — Starting dose 30 mg/m2 given by vein on day 1 of a 21 day cycle.
  Other Names: Taxol
  Arms: Paclitaxel Group
Drug: Sorafenib — Starting dose 200 mg by mouth daily for a 21 day cycle.
  Other Names: Nexavar; BAY 43-9006
  Arms: Sorafenib Group
Drug: Carboplatin — Starting dose AUC 2 by vein on day 1 of a 21 day cycle.
  Other Names: Paraplatin
  Arms: Carboplatin Group

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of bevacizumab (Avastin) and temsirolimus (Torisel) that can be given with 1 of 3 other study drugs --carboplatin (Paraplatin), paclitaxel (Taxol), or sorafenib (Nexavar). The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Temsirolimus is designed to block the growth of cancer cells, which may eventually cause the cancer cells to die.

Carboplatin is designed to damage the DNA (the genetic material of cells)of cancer cells, which may will eventually cause the cancer cells to die.

Paclitaxel is designed to damage the DNA of cancer cells, which may eventually cause the cancer cells to die.

Sorafenib is designed to block the function of important proteins in cancer cells. These proteins, when active, are in part responsible for the abnormal growth and behavior of cancer cells.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, your doctor will decide which study drugs you will receive based on the disease type and on the drugs you have taken in the past.

Every participant will receive bevacizumab and temsirolimus. The study staff will tell you which of the other 3 drugs (carboplatin, paclitaxel, or sorafenib) you will receive.

Once it is decided which drugs you will receive, you will be assigned to a dose level of the drug combination based on when you join this study. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants on each drug combination will receive the lowest doses. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of each dose combination is found.

Your dose of study drugs may be lowered later, if you do not tolerate the study drug combination well.

Once the highest tolerated dose is found for each group, up to 10 more participants will be added to each group at that dose level. This is called an extension group.

Study Drug Administration:

Each cycle is about 21 days or 28 days, depending on which study drug combination you receive.If you experience side effects, the start of the next cycle may be delayed. Your doctor will tell you on which dose level you will be assigned.

SORAFENIB ARM:

If you are assigned to take sorafenib, you will take it by mouth 1 or 2 times every day (the study staff will tell you how often to take it). You should take sorafenib on an empty stomach, either 1 hour before a meal or 2 hours after a meal.

On Day 1 of each cycle, you will receive bevacizumab by vein. The first infusion is over 90 minutes. The next infusion may be over 60 minutes if the first infusion was well-tolerated. If you tolerate the second infusion well, the third infusion may be over 30 minutes.

On Days 1, 8, and 15 of each cycle, you will receive temsirolimus by vein. During Day 1 of Cycle 1, you will receive it over 60 minutes. If you tolerate it well on Day 1 of Cycle 1, it will be given over 30 minutes on Days 8 and 15 of Cycle 1 and over 30 minutes in further cycles, as long you still tolerate it well.

CARBOPLATIN ARM:

If you are assigned to take carboplatin,you will receive it by vein over 1 hour on Day 1 of each cycle.

On Day 1 of each cycle, you will receive bevacizumab by vein. The first infusion is over 90 minutes. The next infusion may be over 60 minutes if the first infusion was well-tolerated. If you tolerate the second infusion well, the third infusion may be over 30 minutes.

On Days 1, 8, and 15 of each cycle, you will receive temsirolimus by vein. During Day 1 of Cycle 1, you will receive it over 60 minutes. If you tolerate it well on Day 1 of Cycle 1, it will be given over 30 minutes on Days 8 and 15 of Cycle 1 and over 30 minutes in further cycles, as long you still tolerate it well.

PACLITAXEL ARM DOSE LEVELS 1-8:

If you are assigned to take paclitaxel on Dose Levels 1 - 8, you will receive it by vein over 3 hours on Days 1, 8, and 15 of each cycle.

On Day 1 of each cycle, you will receive bevacizumab by vein. The first infusion is over 90 minutes. The next infusion may be over 60 minutes if the first infusion was well-tolerated. If you tolerate the second infusion well, the third infusion may be over 30 minutes.

On Days 1, 8, and 15 of each cycle, you will receive temsirolimus by vein. During Day 1 of Cycle 1, you will receive it over 60 minutes. If you tolerate it well on Day 1 of Cycle 1, it will be given over 30 minutes on Days 8 and 15 of Cycle 1 and over 30 minutes in further cycles, as long you still tolerate it well.

PACLITAXEL ARM DOSE LEVELS 9 - 13:

If you are assigned to take paclitaxel on Dose Levels 9 - 13, you will receive paclitaxel by vein over 3 hours on Days 1, 8, and 15 of each cycle.

On Days 1 and 15 of each cycle, you will receive bevacizumab by vein. The first infusion is over 90 minutes. The next infusion may be over 60 minutes if the first infusion was well-tolerated. If you tolerate the second infusion well, the third infusion may be over 30 minutes.

On Days 1, 8, 15, and 22 of each cycle, you will receive temsirolimus by vein. During Day 1 of Cycle 1, you will receive it over 60 minutes. If you tolerate it well on Day 1 of Cycle 1, it will be given over 30 minutes on Days 8, 15, and 22 of Cycle 1 and over 30 minutes in further cycles, as long you still tolerate it well.

Study Visits:

During Cycle 1:

* Urine will be collected for routine tests on Day 1.
* You will have a physical exam, including measurement of your weight and vital signs (blood pressure, breathing rate, heart rate, and temperature).
* You will be asked how well you are able to perform the normal activities of daily living (performance status) on Days 1 and 8.
* Blood (about 1 tablespoon) will be drawn for routine tests on Days 1, 8, and 15.

On Day 1 of Cycles 2 and beyond:

* You will have a physical exam, including of your weight and vital signs..
* Your performance status will be recorded.
* Blood (about 1 tablespoon) and urine will be collected for routine tests

After Cycle 2, you will have a CT scan or MRI scan to check the status of the disease every 2-3 cycles. After 6 months, this may be performed up to every 4 cycles if the doctor thinks it is in your best interest.

Length of Study:

You may remain on study for as long as the doctor thinks it is in you best interest. You will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Bevacizumab, temsirolimus, carboplatin, paclitaxel, and sorafenib are all commercially available. Bevacizumab is FDA approved for the treatment of colorectal cancer and a type of lung cancer. Temsirolimus is FDA approved for the treatment of kidney cancer that has spread. Carboplatin is FDA approved for the treatment of ovarian cancer or non-small cell lung cancer. Paclitaxel is FDA approved for ovarian, breast cancer, and AIDS-related Kaposi's sarcoma. It is also approved in combination with cisplatin for the treatment of ovarian and non-small cell lung cancer. Sorafenib is FDA approved for the treatment of kidney cancer.

The use of these drugs together is investigational.

Up to 278 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion: (For all treatment arms)
2. 1.1 Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that induces a CR rate of at least 10% or improves survival by at least three months.
3. 1.2 Patients must have been off previous chemotherapy or radiotherapy for the three weeks prior to entering this study. Six weeks will be required if the patient has received therapy which is known to have delayed toxicity (mitomycin or a nitrosurea). Five half-lives will be required for biologic/targeted therapies with short (<24 hour) half-lives and pharmacodynamic effects. Patients may have received palliative radiation immediately before (or during) treatment provided radiation does not target the only measurable or evaluable disease.
4. 1.3 Patients must have measurable or evaluable disease
5. 1.4 ECOG performance status </= 2 (Karnofsky >/= 60%, Lansky >/= 50%).
6. 1.5 Patients must have normal organ function defined as: creatinine </= 1.5 x ULN for children and </= 2.0 x ULN for adults; total bilirubin </= 2.0; ALT(SGPT)/AST (SGOT) </= 5 X ULN. In patients with significant liver disease and chronically elevated liver transaminases, ALT/AST may be elevated as high as 8 X ULN.
7. 1.6 Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose.
8. 1.7 Ability to understand and the willingness to sign a written informed consent document.
9. 1.8 Life expectancy of at least 3 months.
10. 1.9 Patients may not be receiving any other experimental agents and/or any other concurrent anticancer agents or therapies except hormonal maintenance.
11. Inclusion: (For carboplatin and paclitaxel arms)
12. 2.1 Patients must have normal marrow function defined as: absolute neutrophil count >/= 1,500/mL; platelets >/= 100,000/mL.
13. 2.2 Patient with neuropathies of CTC grade 1 or less.
14. Inclusion: (For sorafenib arm)
15. 3.1 Patients must have normal marrow function defined as: absolute neutrophil count >/= 1,000/mL; platelets >/= 75,000/mL.

Exclusion Criteria:

1. Exclusion: (For all treatment arms)
2. 4.1 Patients with clinically significant unexplained bleeding within 28 days prior to entering the study.
3. 4.2 Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg on medication).
4. 4.3 Patients with clinically significant cardiovascular disease: History of CVA within 6 months Myocardial infarction or unstable angina within 6 months Unstable angina pectoris New York Heart Association Class > II
5. 4.4 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics on Day 1.
6. 4.5 Pregnant or lactating women.
7. 4.6 History of hypersensitivity to bevacizumab or murine products, temsirolimus or its metabolites, or any component of the formulation.
8. 4.7 Patients with hemorrhagic brain metastases.
9. 4.8 Patients with prior abdominal surgery within 30 days prior to entering the study.
10. 4.9 Medications with potent inducer or inhibitor of P450 3A4 should be avoided within 5 half lives of temsirolimus.
11. Exclusion: (For carboplatin treatment arm)
12. 5.1 Hypersensitivity to carboplatin or any component of the formulation.
13. Exclusion: (For paclitaxel treatment arm)
14. 6.1 Hypersensitivity to paclitaxel or any component of the formulation.
15. Exclusion: (For sorafenib treatment arm)
16. 7.1 History of hypersensitivity to sorafenib or any component of the formulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2010-08-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks
  MTD defined by dose-limiting toxicities (DLTs) that occur during the first four weeks of therapy. DLT defined as any grade 3 or 4 non-hematologic toxicity as defined in NCI CTC v4.0.

SECONDARY OUTCOMES:
Anti-Tumor Efficacy of Temsirolimus and Bevacizumab When Used in Combination with Carboplatin | 56 days
  Anti-tumor efficacy of each drug combination assessed by the WHO criteria if participant has lymphoma.
  Anti-tumor efficacy of each drug combination assessed by the RECIST criteria for all other cancers.
Anti-Tumor Efficacy of Temsirolimus and Bevacizumab When Used in Combination with Paclitaxel | 56 days
  Anti-tumor efficacy of each drug combination assessed by the WHO criteria if participant has lymphoma.
  Anti-tumor efficacy of each drug combination assessed by the RECIST criteria for all other cancers.
Anti-Tumor Efficacy of Temsirolimus and Bevacizumab When Used in Combination with Sorafenib | 56 days
  Anti-tumor efficacy of each drug combination assessed by the WHO criteria if participant has lymphoma.
  Anti-tumor efficacy of each drug combination assessed by the RECIST criteria for all other cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subbiah V, Westin SN, Wang K, Araujo D, Wang WL, Miller VA, Ross JS, Stephens PJ, Palmer GA, Ali SM. Targeted therapy by combined inhibition of the RAF and mTOR kinases in malignant spindle cell neoplasm harboring the KIAA1549-BRAF fusion protein. J Hematol Oncol. 2014 Jan 14;7:8. doi: 10.1186/1756-8722-7-8. PMID 24422672
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org